## Preventing Sexual Violence Through a Comprehensive, Peer-led Initiative NCT03207386 August 19, 2021

## **Data Analyses**

All analyses were estimated in Stata 15. In all analyses, we used multiple imputation (MI; 20 imputed datasets) to address attrition and other missing data (Lang & Little, 2018). To address  $Aim\ 1a$ , we conducted a series of logistic regression analyses, one for each of the dichotomous W3 outcomes (i.e., sexual perpetration, sexual victimization). Covariates were sex (1 = male), ethnicity (1 = Hispanic/Latinx), race (1 = White), sexual orientation  $(1 = sexual\ minority)$ , age (higher = older), school (dummy coded with the largest school as the comparison group), and the W1 outcome score (as applicable to each model).

Data collection protocols allowed for analysis of the long-term impact of the large camp and short-term impact of the small camp. However, because large and small camp attendance (e.g., youth could attend both camps) may co-vary they were included in the same model. That is logistic regression models examined the effects of both large camp attendance ( $0 = did \ not$  attend; 1 = attended) and small camp attendance ( $0 = did \ not \ attend$ ; 1 = attended) on each primary outcome included in the model.